CLINICAL TRIAL: NCT01995578
Title: A Single Arm Phase II Trial of Maintenance Low Dose 5'-Azacitidine Post T Cell Depleted Allogeneic Stem Cell Transplantation for Patients With Myelodysplastic Syndrome and Acute Myelogenous Leukemia With High Risk for Post-Transplant Relapse
Brief Title: Maintenance Low Dose 5'-Azacitidine Post T Cell Depleted Allogeneic Stem Cell Transplantation for Patients With Myelodysplastic Syndrome and Acute Myelogenous Leukemia With High Risk for Post-Transplant Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-192
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-09

CONDITIONS: Myelodysplastic Syndromes (MDS); Acute Myelogenous Leukemia (AML)
Keywords: 5'-Azacitidine; Stem cell transplant; 13-192
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

ARMS (1):
- low dose 5'-azacitidine (Experimental): This is a single arm phase II trial to assess the efficacy and confirm the safety of maintenance therapy with 5'-azacitadine compared to historical control after TCD allogeneic hematopoietic stem cell transplant for patients with MDS and AML who are at high risk of relapse.
  Interventions: Drug: low dose 5'-azacitidine

INTERVENTIONS:
Drug: low dose 5'-azacitidine — 5'-azacitadine will be given at a low dose of 32mg/m2 S.C for 5 days every 28 days (a cycle). Dose de-escalation will be permitted for hematologic and non- hematologic toxicities. Patients will start taking the study drug between days 60-120 post TCD allogeneic hematopoietic stem cell transplant and up to a year post-transplant or until there is a toxicity that requires cessation of therapy. Therefore patients will get between 8-10 cycles. Patients who come off-study for reasons unrelated to toxicities before completing 4 cycles will be replaced Since most cases of relapse occur early post transplant, in the first year, this is the most appropriate time to intervene. Treatment will start as soon as possible.

SUMMARY:
The purpose of this study is to learn if 5'-Azacitidine will help to lower the risk of the disease coming back after a stem cell transplant in patients with MDS and AML. This study will also be looking at the side effects of this medicine.

5'-Azacitidine is an FDA approved drug for treatment of MDS and AML, as well as patients whose disease came back after transplant, where it helped going into remission. It is unclear if 5'-Azacitidine can prevent the disease from coming back after transplant. This study will help show if getting 5'-Azacitidine soon after transplant can lower the risk of your disease coming back.

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone T cell depleted allogeneic hematopoietic stem cell transplantation at MSKCC for:

* De novo myelodysplastic syndromes (MDS): IPSS-1 with poor risk cytogenetics or higher IPSS.
* Acute myelogenous leukemia (AML) in first remission that required more than 1 cycle of treatment to achieve remission or with the following cytogenetic abnormalities: FLT3 mutation, deletion/monosomy of chromosome 5 or 7, MLL gene rearrangement, or more than or equal to 3 cytogenetics abnormalities. Also patients in second or greater remission.
* Patients with Secondary MDS/AML.
* Patients will be considered eligible for the study if after transplant they achieved hematologic (<5% blasts) and cytogenetic remission.
* Patients will be eligible to enter the study between 60-120 days post transplant.
* Age: pediatrics and adults patients - 1 year old-75 years old.
* Karnofsky performance status >=60% for patients >16yo and Lansky performance status >=60% for patients ≤16yo
* Stable blood counts (ANC>1000/uL, Hb>8gr/dL, Plt>50,000/ uL) not supported by transfusions.
* Renal: Serum creatinine <1.5 ULN
* Hepatic: <3xULN ALT and <1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia.
* Cardiac: Adequate cardiac function measured by LVEF>50%. If asymptomatic, pretransplant echocardiogram is adequate. If symptomatic, echocardiogram needs to be repeated.
* Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

Patients will be excluded from the trial if at time of enrollment:

* Active uncontrolled bacterial, fungal or viral infection.
* Evidence of uncontrolled graft-versus-host disease.
* Pulmonary: new onset hypoxia
* Known or suspected hypersensitivity to 5'-azacitadine or mannitol.

  * Evidence of residual disease either by increased blasts count (>5%) or persistence of previous known cytogenetics abnormalities.
* Peripheral blood neutrophil chimerism: less than 95% donor.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roni Tamari, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent and Follow-up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow-up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow-up), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow-up), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Follow-up), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-up), Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose 5'-Azacitidine
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Dose 5'-Azacitidine
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 60 [28 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Relapse Rate
Description: Relapse of MDS or AML will be analyzed as to type and genetic origin of the leukemic cells. These will be defined by morphologic and/or cytogenetic criteria: an increasing number of blasts in the marrow over 5%, by presence of circulating blasts, or by presence of blasts in any extramedullary site as well as presence of previous cytogenetic abnormalities. Other studies assessing for MRD, FACS and FISH assays will be evaluated but would not be considered disease relapse if positive since they are experimental.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 5'-Azacitidine
Number analyzed (Participants) | 32
Participants
  Progression Free | 20
  Complete Response | 2
  Not Entered | 10

2. Secondary Outcome: Overall Survival
Description: Kaplan-Meier methodology will be used to compare overall survival.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 5'-Azacitidine
Number analyzed (Participants) | 32
Participants
  Alive | 20
  Dead | 12

3. Secondary Outcome: Number of Participants Evaluated for Treatment Safety
Description: The safety will be described by tabulating the number of transfusions, frequencies of bleeding and serious infections, and the use of G-CSF support.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 5'-Azacitidine
Number analyzed (Participants) | 32
Participants | 32

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Low Dose 5'-Azacitidine
All-Cause Mortality (participants affected / at risk) | 12/32
Serious Adverse Events (participants affected / at risk) | 10/32
Other Adverse Events (participants affected / at risk) | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose 5'-Azacitidine (N=32)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Intracranial hemorrhage (Nervous system disorders) | 2
Lung infection (Infections and infestations) | 4
Platelet count decreased (Investigations) | 2
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose 5'-Azacitidine (N=32)
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 9
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 5
Anemia (Blood and lymphatic system disorders) | 4
Platelet count decreased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Constipation (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
White blood cell decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT01995578/Prot_SAP_000.pdf